CLINICAL TRIAL: NCT05157061
Title: A Multi-centre, Randomized, Placebo-Controlled, Efficacy Study of Prebiotic Galacto-oligosaccharides on Gastrointestinal Symptom Severity in Patients With Irritable Bowel Syndrome
Brief Title: GOS to Reduce Symptom Severity in IBS
Acronym: EGIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clasado (Industry)
Collaborators: CR2O B.V. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EGIS-01
Record Dates: First submitted 2021-12-01; First posted 2021-12-14 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Irritable Bowel Syndrome; Irritable Bowel Syndrome - Constipation; Irritable Bowel Syndrome - Diarrhoea; Irritable Bowel Syndrome - Mixed
Keywords: Irritable Bowel Syndrome; Diarrhoea; Constipation; Galacto-oligosaccharides (GOS); Symptom severity; Prebiotic; Supplement; Rome IV Criteria
MeSH Terms: conditions — Irritable Bowel Syndrome; Diarrhea; Constipation | interventions — Prebiotics

STUDY DESIGN:
Intervention Model Description: Phase III, randomized, double-blind, placebo-controlled, multi-centre, 8-week intervention study, preceded by a 2-week run-in period, to assess the efficacy of GOS on symptom severity in adult patients with IBS.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study team and DMC are masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GOS arm (Experimental): A single daily dose of a food supplement containing GOS for 8 weeks
  Interventions: Dietary Supplement: Galacto-oligosaccharides (GOS)
- Placebo arm (Placebo Comparator): A single daily dose of maltodextrin, matching in taste, smell, appearance, and solubility, but without active ingredients (i.e. GOS), for 8 weeks
  Interventions: Dietary Supplement: Maltodextrine

INTERVENTIONS:
Dietary Supplement: Galacto-oligosaccharides (GOS) — An 8-week intervention study, preceded by a 2-week run-in period, in which a daily dose of a prebiotic supplement is given to adult patients diagnosed with IBS (diarrhoea, constipation or mixed-type). Patients need to report several symptom experiences and blood and faecal samples are collected.
  Other Names: Prebiotic
  Arms: GOS arm
Dietary Supplement: Maltodextrine — An 8-week intervention study, preceded by a 2-week run-in period, in which a daily dose of a placebo is given to adult patients diagnosed with IBS (diarrhoea, constipation or mixed-type). Patients need to report several symptom experiences and blood and faecal samples are collected.
  Other Names: Placebo
  Arms: Placebo arm

SUMMARY:
IBS is a highly prevalent bowel disorder, characterized by recurrent abdominal pain during bowel movements or a change in bowel habits. Typically, IBS patients experience constipation, diarrhoea or a mix of constipation and diarrhoea, as well as symptoms of abdominal bloating or distension. The chronic and bothersome nature of IBS symptoms negatively affects the quality of life of many patients. Because there are currently limited medical treatment options for IBS, it is important to study new treatments.

IBS can (in part) be caused by an 'imbalance' of the bacteria residing in the intestinal tract. For instance, there may be a lower proportion of specific bacteria that are generally considered beneficial for a persons health. The consumption of non-digestible food ingredients, such as GOS, may stimulate the growth of these beneficial bacteria. GOS is a type of 'prebiotic', which is known to support health and wellbeing of consumers. By restoring the bacterial balance of the intestinal tract, the symptoms of IBS may be reduced after consumption of GOS.

The health effects of the study product (a specific GOS) used in current study was previously investigated in a small group of patients with IBS. Use of the study product indicated a reduction in the patients' symptoms, improvement in the patients' quality of life, and changes in patients' gut bacteria. It is therefore hypothesized that GOS / a specific GOS may reduce the symptom severity of patients with IBS.

This study further evaluates how GOS may improve symptoms of IBS.

DETAILED DESCRIPTION:
A Phase III, randomized, double-blind, placebo-controlled, multi-centre, 8-week intervention study, preceded by a 2-week run-in period, to assess the efficacy of GOS on symptom severity in adult patients with IBS. The study population will consist of 210 adult patients diagnosed in the past 36 months with IBS-Diarrhoea (N =70), IBS-Constipation (N = 70), or IBS-Mixed (N =70).

Irritable bowel syndrome (IBS) is a highly prevalent and multifaceted functional bowel disorder characterized by recurrent abdominal pain associated with defecation or a change in bowel habits in the absence of detectable structural and biochemical abnormalities. Disordered bowel habits are typically present, such as constipation, diarrhoea or a mix of constipation and diarrhoea, as are symptoms of abdominal bloating/distension. The chronic and bothersome nature of IBS symptoms negatively affects patients' quality of life and introduces a substantial economic burden on patients and the healthcare system. The gut microbiota composition and function may play a pivotal role in the pathogenesis of IBS, as a reduction in endogenous bifidobacteria, lactobacilli, and Faecalibacterium prausnitzii concentrations, as well as small bowel bacterial overgrowth have been reported in IBS patients, thereby introducing the gut microbiota as a potential target for treatment and symptom relief. Intervention with non-digestible food ingredients, such as galacto-oligosaccharides (GOS), may form a suitable intervention strategy, as these 'prebiotics' are known to modulate the gastrointestinal (GI) microbiota and support health and wellbeing of the host.

The safety and efficacy of GOS has previously been evaluated in patients with IBS, which demonstrated that GOS may reduce IBS symptom severity, improve quality of life, improve stool consistency and defecation frequency and alter gut microbiota composition, in a safe manner.

As there are currently limited suitable medical treatments for IBS, this study will evaluate the efficacy of GOS in reducing symptom severity of patients with IBS

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have been diagnosed with IBS by a medically trained person/Health Care Professional (HCP).
2. IBS diagnosis to be confirmed according to the Rome-IV criteria by a primary or secondary care clinician, including a gastroenterologist, at study entry
3. An IBS Symptom Severity Scale score of ≥125 points at baseline
4. Male or female between 18 and 64 years of age (age ranges included)
5. Possession of a smartphone
6. Willing and eligible to provide consent and comply with protocol and product intake.

Exclusion Criteria:

1. Unclassifiable IBS (IBS-U) as determined by Investigator
2. Use of products marketed as prebiotics, probiotics or synbiotics within 4 weeks prior to study entry (e.g. Yakult, Actimel, Activia, VSL#3, Kefir).

   o Regular cheese or yogurt containing lactic acid bacteria are not an exclusion criterion.
3. Systemic antibiotic or antimycotic treatment within 4 weeks prior to study entry
4. Use of laxatives or antidiarrheal medication within 1 week prior to study entry
5. An unstable antidepressant/antipsychotic treatment regimen within 3 months prior to study entry (i.e. treatment should be stable for at least 3 months prior to study entry).
6. Confirmed lactose intolerance, defined as patients who report response to dietary elimination of lactose/dairy products. Confirmation is patient-reported and not done within the scope of this study.
7. Confirmed food allergy, with reported confirmation based on OFC, IgE, or skin prick test. Confirmation is patient-reported and not done within the scope of this study.
8. Galactosemia (galactose metabolism disorder)
9. Following diets likely to affect study outcomes, including:

   o low FODMAP, KETO/high-fat, gluten free/coeliac, paleo, weight loss, caloric restriction, low-carb, 5:2/whole day energy restriction, Atkins/high-protein, sugar-free, single-food, juicing/any day of juicing, any other restriction diet (e.g. very low calory), or vegan diets (GOS is derived from cow's milk).
10. Severe illness(es) or medical condition(s), including gastrointestinal pathologies:

    o GI ulcers, coeliac disease, inflammatory bowel disease, bowel cancer, bowel resection, , bariatric surgery, acute or chronic diarrhoea secondary to confirmed infectious gastroenteritis, or enteral or parenteral nutrition.
11. Subjects suffering from auto-immune disorders (e.g. Rheumatoid Arthritis, Systemic lupus erythematosus, Multiple Sclerosis, Graves' Disease) that require treatment with an immune modulator treatment or anti-inflammatory medication
12. Surgical operations to the mouth or gastrointestinal tract within 4 weeks prior to study entry, or planned during the study

    o Appendectomy within 6 months prior to study entry
13. Recent unintended weight loss:

    o >5% of total body weight within 6 months prior to study entry
14. Excessive alcohol consumption (>14 units per week) and/or drug abuse
15. Pregnancy and lactation, or plan to become pregnant during the study period
16. Participation in other studies involving investigational or marketed products concomitantly or within 3 months prior to study entry
17. Changes in diet, supplement or medication use likely to affect study outcomes (i.e. medication that influences GI function) within 4 weeks prior to study entry or planned during the study (at the discretion of the Investigator). For example, the following medications will influence GI function and changes must be avoided: opioids, prokinetics (domperidone, metoclopramide, prucalopride), antispasmodics (peppermint oil, buscopan), and acid suppressants (PPI, H2 blockers). Of note: the intake of fibres (e.g. psyllium husk) may be used provided that the participant has been using this as a supplement for more than 4 weeks prior to study participation and intake does not change during the course of participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2021-10-26 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2024-08-06 (Actual)

PRIMARY OUTCOMES:
IBS symptom Severity | Baseline to end of the study (Day 56).
  The difference in total IBS symptom severity between treatment arms as measured by mean composite IBS Symptom Severity Scale scores. The IBS System Severity Scores Scale consists of 5 questions each with scales ranging from 0 to 100, divided into steps of 10, whereby a score of 0 reflects the best outcome, and a score of 100 reflects the worst outcome.

SECONDARY OUTCOMES:
Abdominal pain | During the intervention period (8 weeks)
  The difference in abdominal pain between treatment groups as measured by the mean abdominal pain symptom scores as reported by patients in their electronic diaries. Patients are requested to rate their worst abdominal pain over the past 24 hours on a scale from 0 = no abdominal pain, 10 = worst possible abdominal pain.
Bloating. | During the intervention period (8 weeks)
  The difference in bloating between treatment groups as measured by the mean bloating symptom scores as reported by patients in their electronic diaries. Patients are requested to to rate their worst bloating symptoms over the past 24 hours, on a scale from 0 = no bloating, 10 = worst possible bloating.
Global IBS improvement | During the intervention period (8 weeks)
  The difference in global IBS improvement between treatment arms as measured by the mean IBS Global Improvement Scale scores. Patients are requested to rate their IBS signs or symptoms overall over the past 7 days on a scale from 1 = significantly relieved to 7 = significantly worse.
Stool consistency | During the intervention period (8 weeks)
  The difference in stool consistency between treatment arms, per subtype of IBS**, as measured by the median Bristol Stool Form Scale stool type. The Bristol Stool Form Scale stool types vary from 1 (separate hard lumps) to 7 (watery, no hard pieces). Normal stools would be rated in the middle of this scale (3, 4, or 5)
Defecation frequency | During the intervention period (8 weeks)
  The difference in defecation frequency between treatment arms, per subtype of IBS**, as measured by the mean patient-reported defecation frequency.
Quality of Life IBS-QOL score | At the end of the study (Day 56)
  The difference in quality of life between treatment arms as measured by the mean composite IBS Quality of Life scores. The IBS Quality of Life validated questionnaire offers patients 34 statements concerning bowel problems (Irritable Bowel Syndrome, IBS) and how these affected the patient over the past 30 days, Scores range from 1 (not at all) to 5 (extremely)
Anxiety and depression | At the end of the study (Day 56)
  The difference in anxiety and depression between treatment arms, evaluated separately using the mean IBS Hospital Anxiety and Depression Scale scores. The Hospital Anxiety and Depression scale asks patients to rate how they feel in 14 questions, each offering 4 different outcomes ranging from the best possible feeling to worst possible feeling
Nature, incidence, frequency, severity of adverse events/serious adverse events and relationship to the study intervention. | During the intervention period (8 weeks)
  To assess the safety of treatment with GOS in patients with IBS
Rescue medication | From screening to end of intervention period (10 weeks)
  Difference in use of rescue medication between treatment arms

OTHER OUTCOMES:
Immune function | At the end of the study (Day 56).
  The difference in immune function between treatment arms as determined by blood markers of immune function.
Gut microbiome composition | At the end of the study (Day 56).
  The difference in gut microbiome composition between treatment arms as determined by faecal metagenomics.
Blood metabolites | At the end of the study (Day 56).
  The difference in blood metabolites between treatment arms as determined by blood metabolomic analysis.
Correlation between blood metabolites and gut microbiome | At the end of the study (Day 56).
  The correlation of blood metabolites and gut microbiome in both treatment arms, and the difference between arms.
Correlation between gut microbiome and mean composite IBS-Symptom Severity Scores | At the end of the study (Day 56).
  The correlation of gut microbiome and mean composite IBS-Symptom Severity Scores in both treatment arms, and the difference between arms.

CONTACTS AND LOCATIONS:
Overall Officials: Lucien F. Harthoorn, PhD., Study Director — Clasado Research Services Limited
Locations (9):
- University Hospital Leuven location Gasthuisberg, Leuven, Belgium
- Netherlands (3):
  - Jeroen Bosch Ziekenhuis, Gastroenterology department, 's-Hertogenbosch, North Brabant
  - Medisch Centrum Leeuwarden (MCL), Leeuwarden, Provincie Friesland
  - Ziekenhuis Gelderse Vallei, Afdeling Maag-Darm-Leverziekten, Ede
- United Kingdom (5):
  - Leeds Teaching Hospital NHS Trust in association with the University of Leeds, Leeds, North Yorkshire
  - County Durham &Darlington NHS Foundation trust, University Hospital of North Durham, Durham
  - Barts Health NHS Trust, Wingate Clinical Trials Facility, London
  - Manchester University NHS Foundation Trust, Wythenshawe Hospital, Neurogastroenterology Unit, Manchester
  - NIHR National Patient Recruitment Centre Newcastle, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No